CLINICAL TRIAL: NCT03735797
Title: Cancer Stem Cells in Acute Leukemia
Status: Active, not recruiting | Type: Observational
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Other Study IDs: SH Can Stem
Record Dates: First submitted 2018-07-26; First posted 2018-11-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bone marrow aspirate or peripheral blood sample collection — Collection of specimen samples only

SUMMARY:
Descriptive study of acute leukemia patients. Bone marrow aspirate or peripheral blood samples will be analyzed by next-generation sequencing for novel gene signatures and variations in transcriptional and epigenetic regulatory elements such as ARID5B and SALL4 variants.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or relapsed acute leukemia (AML or ALL)
* Plan to undergo diagnostic bone marrow aspirate or peripheral blood if clinically indicated (i.e. WBC>50,000 and bone marrow contraindicated)
* Age 1 month to 30 years
* Understand and provide informed consent (subject if>18, legal guardian if<18)

Exclusion Criteria:

* Age 0 to 4 weeks
* Treatment related leukemia or leukemia secondary to MDS
* Situations that would limit compliance with study requirements or ability to willingly give consent

Ages: 1 Month to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study team will enroll approximately 50 subjects (age 1 month to 30 years) with newly diagnosed or relapsed acute leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-07-12 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
ARID5B polymorphism/mutation status | 5 years
  Correlation of our experimentally validated Arid5b dependent transcriptional signature with primary patient samples measured by patient ARID5B expression and polymorphisms.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanford, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No